CLINICAL TRIAL: NCT03694327
Title: Clinical Trial of an Innovative Digital Therapeutic for Smoking Cessation With Biochemical Verification
Brief Title: Innovative Digital Therapeutic for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: My Digital Study (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT-101-002
Record Dates: First submitted 2018-09-12; First posted 2018-10-03 (Actual); Results first posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-05

CONDITIONS: Smoking Cessation; Nicotine Addiction; Drug Addiction; Drug Dependence; Tobacco Dependence; Tobacco Use Disorder; Substance Use Disorder; Tobacco Smoking
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder; Substance-Related Disorders; Tobacco Smoking

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment A Mobile Application (Experimental): Treatment A Digital Intervention: Smartphone application designed to assist with smoking cessation.
  Interventions: Device: CT-101-M
- Treatment B Mobile Application (Active Comparator): Treatment B Digital Intervention: Smartphone application designed to assist with smoking cessation.
  Interventions: Device: QuitGuide

INTERVENTIONS:
Device: CT-101-M — Mobile Application
  Arms: Treatment A Mobile Application
Device: QuitGuide — Mobile Application
  Arms: Treatment B Mobile Application

SUMMARY:
This study is comparing the efficacy of two smoking cessation apps.

DETAILED DESCRIPTION:
Given that tobacco smoking is the leading cause of preventable death in the US, the development of effective cessation programs is critical; mobile phone applications represent a novel, accessible platform for helping smokers quit. This research project seeks to compare the efficacy of two smoking cessation apps. In a blinded, randomized, controlled study, current smokers motivated to quit will use a smoking cessation app for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 to 65
* Fluent in written and spoken English (confirmed by ability to read and comprehend Informed Consent Form)
* Lives in the United States
* Smokes at least 5 cigarettes daily
* Is interested in quitting in the next 30 days
* The participant owns and has access to an iPhone with iOS 9 or greater capabilities, or an Android with OS 7 or greater capabilities
* The participant is willing and able to receive SMS text messages on their smartphone
* The participant is willing and able to receive email messages.
* Ability to confirm download of installed treatment arm app via telephone on randomization date.
* One half of the study sample will be recruited from the general population of smokers via social media advertisements
* One half of the study sample will be recruited via mail form a Magellan Behavioral Health value-based care network

Exclusion Criteria:

* Prior use of Treatment A Digital Intervention or Treatment B Digital Intervention
* Current use of pharmacotherapy for smoking cessation or nicotine replacement therapy (NRT)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Iacoviello, PhD, Principal Investigator — My Digital Study
Locations (1):
- My Digital Study, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment A Mobile Application: Treatment A Digital Intervention: Smartphone application designed to assist with smoking cessation.
  CT-101-M (Mobile Application): A reduced-functionality minimal viable product (MVP) version of Clickotine (CT-101).
Period: Overall Study
Arm/Group | Treatment A Mobile Application | Treatment B Mobile Application
Started | 79 | 79
Completed | 66 | 56
Not Completed | 13 | 23
Not completed — Lost to Follow-up | 13 | 23

BASELINE CHARACTERISTICS:
Population: The population enrolled was US only, male or female, ages 18 to 65, and smoke at least 5 cigarettes per day with an interest in quitting smoking within the next 30 days. Participants enrolled had not used Clickotine or QuitGuide; and were not using an NRT at the time of enrollment.
Groups:
- Treatment A Mobile Application (CT-101-M): Treatment A Digital Intervention: Smartphone application designed to assist with smoking cessation.
  CT-101-M (Mobile Application): A reduced-functionality minimal viable product (MVP) version of Clickotine (CT-101).
- Treatment B Mobile Application (QuitGuide): Treatment B Digital Intervention: Smartphone application designed to assist with smoking cessation.
  QuitGuide: Mobile Application
- Total: Total of all reporting groups
Arm/Group | Treatment A Mobile Application (CT-101-M) | Treatment B Mobile Application (QuitGuide) | Total
Number analyzed (Participants) | 79 | 79 | 158
Age, Customized [Count of Participants; unit: Participants] — Measured via Self-Report in the Baseline Survey.
  Participants
    18-39 years | 60 | 59 | 119
    40-59 years | 18 | 19 | 37
    60+ years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Measured via Self-Report in the Baseline Survey.
  Participants
    Female | 52 | 55 | 107
    Male | 27 | 24 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Measured via Self-Report in the Baseline Survey.
  Participants
    White | 59 | 65 | 124
    All Other Races | 20 | 14 | 34
Region of Enrollment [Count of Participants; unit: Participants] — Measured via Self-Report in the Baseline Survey.
  Participants
    United States | 79 | 79 | 158
Family Size, Categorical [Count of Participants; unit: Participants] — Measured via Self-Report in the Baseline Survey.
  Participants
    0-2 | 31 | 32 | 63
    3-5 | 47 | 40 | 87
    6+ | 1 | 7 | 8
Education, Categorical [Number; unit: participants] — Measured via Self-Report in the Baseline Survey.
  participants
    < HS or GED | 17 | 12 | 29
    High School | 10 | 13 | 23
    > High School | 52 | 54 | 106
Income Range, Categorical [Count of Participants; unit: Participants] — Measured via Self-Report in the Baseline Survey.
  Participants
    Less than $20,000 | 16 | 21 | 37
    $20,000 to $55,000 | 38 | 38 | 76
    $55,000 to $100,000 | 15 | 13 | 28
    Over $100,000 | 10 | 7 | 17
Internet Frequency, Categorical [Count of Participants; unit: Participants] — Measured via Self-Report in the Baseline Survey.
  Participants
    A few times per day | 3 | 1 | 4
    At least once per day but less than several times | 3 | 4 | 7
    At least several times per day | 32 | 33 | 65
    Several times per day | 41 | 41 | 82
Fagerstrom Test for Nicotine Dependence [Count of Participants; unit: Participants] — The Fagerstrom Test for Nicotine Dependence is a standard instrument for assessing the intensity of physical addiction to nicotine. The test was designed to provide an ordinal measure of nicotine dependence related to cigarette smoking. In scoring the Fagerstrom Nicotine Dependency Test, yes/no items are scored from 0 to 1 and multiple-choice items are scored from 0 to 3. The items are added to yield a total score of 0-10. The higher total Fagerstrom score indicates a more intense/ higher dependency to nicotine (Heatherton, et. al, 1991)
  Participants
    0-3 | 21 | 19 | 40
    4-7 | 48 | 52 | 100
    8+ | 10 | 8 | 18
Money Spent on Cigarettes (Per Month) [Count of Participants; unit: Participants] — Measured via Self-Report in the Baseline Survey.
  Participants
    Less than $15 | 4 | 9 | 13
    $16 to $30 | 27 | 23 | 50
    $31 to $50 | 33 | 33 | 66
    More than $50 | 15 | 14 | 29
Quit Duration [Count of Participants; unit: Participants] — Participants longest prior quit attempt was measured via self-report in the Baseline Survey.
  Participants
    Less than a week | 13 | 19 | 32
    1 week to 1 month | 18 | 17 | 35
    1 month to 6 months | 23 | 22 | 45
    6 months to 1 year | 15 | 13 | 28
    More than 1 year | 7 | 6 | 13
    N/A | 3 | 2 | 5
Prior Quit Attempts [Count of Participants; unit: Participants] — Participants prior quit attempts were measured via self-report in the Baseline Survey.
  Participants
    0 | 5 | 5 | 10
    1 | 12 | 19 | 31
    2 | 16 | 20 | 36
    3 | 17 | 11 | 28
    4 | 6 | 12 | 18
    5 | 12 | 4 | 16
    N/A | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: 30-Day Sustained Abstinence From Smoking
Description: Self-reported abstinence from smoking was assessed in the 8-Week Outcome Survey.
Time Frame: Upon completion of 8-week period
Population: The study population was randomized 1:1 across Treatment A (CT-101-M) and Treatment B (QuitGuide). The population enrolled was US only, male or female, ages 18 to 65, and smoke at least 5 cigarettes per day with an interest in quitting smoking within the next 30 days. Participants enrolled had not used Clickotine or QuitGuide; and were not using an NRT at the time of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A Mobile Application (CT-101-M) | Treatment B Mobile Application (QuitGuide)
Number analyzed (Participants) | 79 | 79
Participants
  Reported Smoking in the Last 30 Days | 69 | 66
  Reported Not Smoking in the Last 30 Days | 10 | 13

2. Secondary Outcome: Feasibility of Biochemical Verification of Smoking Cessation
Description: Confirmation with the remote CO assessment was conducted to assess concordance between self-report and remote CO assessment results. Abstinence as per the CO assessment was defined as an iCO reading of fewer than 7ppm exhaled CO.
Time Frame: Upon completion of 8-week period
Measure: Mean (Standard Deviation); unit: PPM
Arm/Group | Treatment A Mobile Application (CT-101-M) | Treatment B Mobile Application (QuitGuide)
Number analyzed (Participants) | 47 | 46
PPM | 9.766 (11.099) | 8.609 (9.448)

3. Secondary Outcome: NRT and Smoking Cessation Pharmacotherapy Use
Description: Self-reported NRT and smoking cessation pharmacotherapy use will be acquired via the outcome survey. Cessation rates will be compared between those using/not using pharmacotherapy.
Time Frame: Upon completion of 8-week period
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A Mobile Application (CT-101-M) | Treatment B Mobile Application (QuitGuide)
Number analyzed (Participants) | 79 | 79
Participants
  Used NRT (or other pharmaceutical quit aids) | 10 | 15
  Did not Use NRT (or other pharmaceutical quit aids) | 56 | 41
  Not Reported | 13 | 23

ADVERSE EVENTS:
Time Frame: AE collection occurred 8 weeks after participant began treatment.
Description: Adverse event and serious adverse event definitions used are the same as clinilcaltrials.gov.
  Method of collection: Participants were instructed to contact the study coordinator via a study-specific e-mail and phone number in the event they experienced any adverse event during their participation in the study.
Arm/Group | Treatment A Mobile Application (CT-101-M) | Treatment B Mobile Application (QuitGuide)
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/79 | 1/79
Other Adverse Events (participants affected / at risk) | 11/79 | 5/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A Mobile Application (CT-101-M) (N=79) | Treatment B Mobile Application (QuitGuide) (N=79)
Diabetic Ketoacidosis (Endocrine disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A Mobile Application (CT-101-M) (N=79) | Treatment B Mobile Application (QuitGuide) (N=79)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection Viral NOS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Concussion with no loss of consciousness (General disorders) | 1 (1) | 0 (0)
Fractured Coccyx (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Borderline Personality (Psychiatric disorders) | 1 (1) | 0 (0)
Acute Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Knee Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT03694327/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT03694327/SAP_001.pdf